CLINICAL TRIAL: NCT00182533
Title: Sertraline in the Treatment of Generalized Social Phobia With Comorbidity
Brief Title: Sertraline in Generalized Social Phobia With Co-Occurring Anxiety and Mood Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study drug could not be re-supplied
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02-195
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2017-03

CONDITIONS: Phobia, Social; Panic Disorder; Agoraphobia; Obsessive-Compulsive Disorder; Anxiety Disorders; Major Depressive Disorder
Keywords: Generalized social phobia; Comorbid panic disorder with agoraphobia; Comorbid obsessive compulsive disorder; Comorbid generalized anxiety disorder; Comorbid major depressive disorder/Dysthymia
MeSH Terms: conditions — Phobia, Social; Panic Disorder; Agoraphobia; Obsessive-Compulsive Disorder; Anxiety Disorders; Depressive Disorder, Major; Dysthymic Disorder | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sertraline
  Interventions: Drug: Sertraline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — 25 - 200 mg/day x 16 weeks
  Other Names: Zoloft
  Arms: 1
Drug: Placebo — 25 - 200 mg/day x 16 weeks
  Arms: 2

SUMMARY:
Selective serotonin reuptake inhibitors (SSRIs) including sertraline have been found to be effective in the treatment of generalized social phobia (GSP). However, virtually all of the current treatment studies with medicines, including the SSRIs, have excluded patients with social phobia who have other co-occurring conditions. In fact, 80% of individuals suffering with primary social phobia have at least one other anxiety. This study will evaluate the safety and efficacy of sertraline in the treatment of generalized social phobia with co-occurring anxiety and mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with primary Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) GSP plus at least one of the following comorbid DSM-IV anxiety disorders:

  * panic disorder with agoraphobia
  * obsessive compulsive disorder
  * major depressive disorder
  * generalized anxiety disorder
* Score on LSAS > 50
* Score on MADRS < 25

Exclusion Criteria:

* Any other primary AXIS-I diagnosis
* Criteria for alcohol/substance abuse/dependence
* History (Hx) of bipolar disorder, schizophrenia or other psychotic disorder
* A comorbid Axis II cluster A personality disorder
* Current increased risk of concomitant suicide
* Allergy/previous intolerance during an adequate trial (50mg/day for minimum of 4 weeks) of sertraline
* Participation in any clinical trial 30 days prior to entering the study
* Unable to tolerate being free of/shows signs of withdrawal from benzodiazepines for 4 weeks
* Hx of seizures
* Thyroid problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2002-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression - Improvement ≤ 2 | 16 weeks
Liebowitz Social Anxiety Scale [LSAS] (mean change from baseline) | 16 weeks

SECONDARY OUTCOMES:
Mean change from baseline on the following scales: Quality of Life and Employment Satisfaction Questionnaire | 16 weeks
Sheehan Disability Scale | 16 weeks
Social Phobia Scale | 16 weeks
Brief Social Phobia Scale | 16 weeks
Penn State Worry Questionnaire | 16 weeks
Panic and Agoraphobia Scale | 16 weeks
Davidson Trauma Scale | 16 weeks
Social Anxiety Spectrum Self-Report (SHY-SR) | 16 weeks
Yale-Brown Obsessive Compulsive Scale | 16 weeks
Montgomery-Asberg Depression Rating Scale (MADRS) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada